CLINICAL TRIAL: NCT00708188
Title: Evaluation of Multidetector Raw Computerized Tomography in the Etiological Analysis of Acute Ischemic Stroke: the "COCASE" Protocol.
Brief Title: Multidetector Raw CT as a Single Tool in the Setting of Ischemic Stroke
Acronym: COCASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006.431/24
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2013-07

CONDITIONS: Ischemic Stroke
Keywords: Stroke, ischemic, etiology, TOAST, CT, multidetector
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multidetector raw CT (Experimental)
  Interventions: Device: Multidetector raw CT

INTERVENTIONS:
Device: Multidetector raw CT — Multidetector raw CT

SUMMARY:
This is a prospective study including acute ischemic stroke patients aged 18 to 90. Multidetector raw CT is performed in acute ischemic stroke patients. Heart, neck vessels and brain arteries are studied during the same acquisition. Results are compared with the standard methods including transesophageal echocardiography (TEE), Doppler ultrasound (DUS) and MR angiography (MRA) of neck vessels. The main criteria is the ability of CT to classify the stroke etiology correctly according to the TOAST classification in comparison with the standard methods.

ELIGIBILITY:
Inclusion Criteria:

* Acute (< 1 week) ischemic stroke patient aged 18 to 90
* Informed consent obtained
* Presence of health insurance

Exclusion Criteria:

* Pregnancy or absence of efficient contraceptive method
* Allergy
* Allergy to contrast material
* Asthma
* Renal failure (blood creatinine > 130 µmoles/l, creatinine clearance < 80 ml/mn according to Cockroft method)
* Myeloma
* Hyperthyroidism (uncontrolled)
* Difficulties to synchronize CT to heart rhythm
* Contra-indication to TEE or MRI
* Absence or retirement of informed consent
* Absence of health insurance

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Ability of CT to classify the stroke etiology correctly (TOAST classification) in comparison to reference methods (MRA, DUS, TEE) | classify the stroke etiology

SECONDARY OUTCOMES:
Ability of CT to detect the source of stroke in each etiological group. Reliability of CT in quantitative measures of artery stenosis, aortic atheroma, heart thrombus, heart tumors). Tolerance of CT | detect the source of stroke

CONTACTS AND LOCATIONS:
Overall Officials: DOUEK Philippe, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Cardiologique Louis Pradel, Bron, France

REFERENCES:
- [Result] Boussel L, Cakmak S, Wintermark M, Nighoghossian N, Loffroy R, Coulon P, Derex L, Cho TH, Douek PC. Ischemic stroke: etiologic work-up with multidetector CT of heart and extra- and intracranial arteries. Radiology. 2011 Jan;258(1):206-12. doi: 10.1148/radiol.10100804. Epub 2010 Nov 9. PMID 21062925